CLINICAL TRIAL: NCT02879422
Title: Study of the Association Between Genetic Markers (Endothelial Lipase and Aldose Reductase) and Proliferative Diabetic Retinopathy
Brief Title: Genetic Markers and Proliferative Diabetic Retinopathy
Acronym: REDIAGEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PR12040
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2021-02

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — Genetic Testing

ARMS (2):
- Diabetic patients with proliferative diabetic retinopathy (Other)
  Interventions: Genetic: genetic analysis
- Diabetic patients with non proliferative diabetic retinopathy (Other)
  Interventions: Genetic: genetic analysis

INTERVENTIONS:
Genetic: genetic analysis

SUMMARY:
Type 2 Diabetes (TD2) is the leading cause of new cases of preventable blindness in these countries (and the gold-standard treatment, laser photocoagulation has proven to be effective in preventing vision loss at the end stage of eye disease due to proliferative diabetic retinopathy (PDR) that occurs in 3 to 6 % of the cases.Therefore, the ongoing search for predictive factors of sight threatening stages of diabetic retinopathy has become more important.

Previous studies that have examined candidate predictive factors for diabetic eye disease have mostly focused on systemic risk factors leading to PDR. Among various clinical parameters, increased HbA1c % levels, uncontrolled blood pressure, diabetes duration, neuropathy and elevated triglycerides have been associated with PDR.

Some genetic factors may also account for the development of PDR and are prospectively considered in this study .

DETAILED DESCRIPTION:
In a previous study (2011), investigators demonstrated a statistically significant relation between the Endothelial Lipase(EL) c.584C>T polymorphism and the occurrence of diabetic retinopathy in 396 french patients with diabetes type 2 (DT2) with a longitudinal follow-up.

Secondly (2014) in a subgroup of 287 DT2 patients, investigators showed the impact of the EL rare T allele was consistent with a recessive mode of inheritance, with homozygotes for the rare allele differing from the carriers of the major allele. Importantly, the homozygotes for the rare T allele were more likely to present with advanced stages of diabetic retinopathy (severe non proliferative and proliferative disease) and particularly with proliferative diabetic retinopathy (PDR).

Based on this model investigators decided to conduct a case-control prospective study comparing 155 french patients with DT2 with PDR (cases) and 155 french patients with DT2 without PDR (controls) on the basis of two genetic parameters: EL c.584C>T polymorphism that investigators previously studied and the C(-106)T aldose reductase polymorphism widely studied in diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients
* patient with proliferative diabetic retinopathy (for arm 1)
* patient with non proliferative diabetic retinopathy (for arm 2)
* patient older than 18 years
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Proliferative retinopathy diabetic | Day 0
  diabetic retinopathy with a preretinal and / or prepapillary neovascularization diagnosed using ultra-wide-field imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Result] Henry A, Boigelot T, Moura TF, Leclercq I, Barbe C, Thiery A, Djerada Z, Nazeyrollas P, Clavel C, Cornillet-Lefebvre P, Berrod JP, Creuzot-Garcher C, Meyer L, Gaucher D, Guerci B, Lenoble P, Milazzo S, Perone JM, Arndt C, Durlach V. No association of endothelial lipase and aldose reductase polymorphisms with proliferative diabetic retinopathy: Results of the French prospective multicenter REDIAGEN study. Diabetes Metab. 2024 May;50(3):101533. doi: 10.1016/j.diabet.2024.101533. Epub 2024 Apr 1. No abstract available. PMID 38570135